CLINICAL TRIAL: NCT04055467
Title: Brain Imaging of Nicotinic Acetylcholine Receptors in Tobacco Users and Nonusers
Brief Title: Brain Imaging in Tobacco Smokers During a Quit Attempt
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00173536; 1R21DA047795-01A1 (NIH)
Record Dates: First submitted 2019-08-12; First posted 2019-08-13 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Tobacco Use Disorder; Tobacco Smoking
Keywords: smoking cessation; neuroimaging; nicotinic acetylcholine receptors; abstinence
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking; Smoking Cessation | interventions — 3-(1,4-diazabicyclo(3.2.2)nonan-4-yl)-6-fluorodibenzo(b,d)thiophene 5,5-dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [F18]-ASEM + Contingency Management (Other): PET radiopharmaceutical 3-(1,4-diazabicyclo[3.2.2]nonan-4-yl)-6 [18F]fluorodibenzo[b,d]thiophene 5,5-dioxide with incentive payments.
  Interventions: Drug: [F18]-ASEM (3-(1,4-diazabicyclo[3.2.2]nonan-4-yl)-6-[18F]fluorodibenzo[b,d]thiophene 5,5-dioxide); Behavioral: Contingency Management

INTERVENTIONS:
Drug: [F18]-ASEM (3-(1,4-diazabicyclo[3.2.2]nonan-4-yl)-6-[18F]fluorodibenzo[b,d]thiophene 5,5-dioxide) — Brain imaging of alpha-7 nicotinic acetylcholine receptors
  Other Names: [F18]-ASEM
Behavioral: Contingency Management — Incentive payments contingent upon provision of samples that meet criterion levels of exhaled carbon oxide and urinary cotinine at study visits
  Other Names: Incentive payments

SUMMARY:
The proposed study will help fill gaps in existing research by determining if nicotine-dependent cigarette smokers show changes in α7 nicotinic acetylcholine receptor (nAChR) availability when compared to matched historical controls using positron emission tomography (PET) imaging and the radioactive ligand [18F]-ASEM (3-(1,4-diazabicyclo[3.2.2]nonan-4-yl)-6 [18F]fluorodibenzo[b,d]thiophene 5,5-dioxide), an α7 nAChR antagonist. The study will also explore whether α7 nAChR availability influences clinically relevant measures of tobacco abstinence (e.g., withdrawal and craving, cognitive impairment), self-reported cigarettes per day, and time to relapse during an 8-day quit attempt during which smokers can receive escalating payments contingent upon providing objective evidence (breath CO and urinary cotinine) of smoking abstinence.

DETAILED DESCRIPTION:
The primary objective of this basic clinical research study is to examine the role of the alpha7-nicotinic acetylcholine receptors (nAChRs) in tobacco use disorder. nAChRs are the primary site of action for nicotine (the main psychoactive component of tobacco). The most common types of nAChRs are heteromeric nAChRs containing beta2 subunits and homomeric nAChRs, which contain only alpha7 subunits. It is currently unknown if or how chronic tobacco use affects alpha7 nAChR in humans. The investigators' working hypothesis is brain alpha7 nAChR density associated with chronic nicotine exposure and the development of tobacco use disorder may be influence severity of tobacco craving and withdrawal during early smoking abstinence.

Proposed group sample sizes are 18 tobacco smokers (accrual) and 18 nonsmokers (drawn from historical and contemporary controls in ongoing studies). Media-recruited male and female heavy smokers will be assessed for study inclusion/exclusion criteria using a structured diagnostic interview and a standard battery of instruments, as well as a medical exam to determine general health. Study candidates also provide breath and urine samples to determine biomarkers of tobacco use (breath carbon oxide and urinary cotinine levels), other drug use (breath alcohol and urine toxicology) and for females a pregnancy test. To ensure there are a sufficient number of subjects, 60 subjects will be screened for study eligibility and assessed for matching criteria (age, race and sex). Groups (smokers vs. non-smokers) will include equal numbers of males and females. In addition, male and female smokers will be matched for tobacco use disorder severity using symptom counts (DSM 5).

Eligible subjects will be enrolled in an outpatient protocol completed at the Behavioral Pharmacology Research Unit (BPRU) at the Johns Hopkins Bayview Medical Center, and at the Johns Hopkins Hospital (JHH) PET imaging Center. Abstinent smokers (as verified by CO and cotinine, see below) will complete an magnetic resonance imaging (MRI) scan and a PET scan with the alpha-7 nAChR radiotracer [18F]-ASEM. Matched historical controls will have completed the MRI and PET scans previously.

Tobacco users will receive contingency management incentive payments for verified smoking abstinence (Intervention 2, behavioral counseling). Smokers will continue in the study after the PET scan and complete an 8-day practice quit attempt. To evaluate smoking abstinence and lapse behavior, smokers will be asked to complete study six visits with a practice quit attempt. Smoker will receive the incentive intervention for smoking abstinence. At each visit, smokers will provide carbon monoxide (CO) and urine samples, and complete assessment instruments to self-report on daily symptoms of nicotine withdrawal and craving, and number of cigarettes smoked. The incentive intervention is a validated, established intervention for smoking cessation. At each visit, smokers will receive escalating incentive payments contingent upon provision of samples that meet study defined abstinence criteria. The incentive earning schedule starts at $9 on day 1 of abstinence and increases by $1.50 for each day of verified abstinence to $19.50 on day 8. To boost the incentive for abstinence, provision of samples that meet bonus abstinence (cotinine <100 ng/ml day 8) results additional $10 or $20 bonus payments. The incentive earnings schedule includes allowance for a slip, and a reset contingency to allow smokers to retry the quit attempt and complete the study. This incentive earnings schedule with resets is of high magnitude to reinforce abstinence, and increase participant retainment. The number of days in the quit attempt (8) yields a sufficient sample to examine both withdrawal and biomarkers (CO and cotinine) to quantify number of days in which use of any nicotine occurred vs. days participants were compliant in maintaining abstinence. These data will be utilized to explore the relationship of alpha7-nAChR availability to these clinically meaningful measures of tobacco use and abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be healthy volunteers
* Regular tobacco smokers for a period of 2 or more years
* Positive breath carbon monoxide (CO)
* Cotinine positive urine test
* Meet DSM-V criteria for tobacco use disorder.

Exclusion Criteria:

* Meets DSM-5 criteria for alcohol use disorder or substance use disorder (excluding tobacco use disorder)
* Meets DSM-5 Psychiatric Disorder; in or in need of treatment
* History of seizures, seizure disorder or closed head trauma
* HIV positive
* Weight > 350 lbs
* < 5th grade reading level
* Recent use of smoking cessation products
* If female: pregnant, lactating, planning pregnancy; positive urine pregnancy screen
* Any condition which would preclude MRI
* Radiation exposure in the last year that when combined with the study protocol would exceed the annual limits.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise Weerts, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Elise Weerts, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tobacco Smokers During a Quit Attempt: Abstinent tobacco smokers receive a MRI and a PET scan with the alpha7-nAChR radiotracer [18F]-ASEM to assess alpha-7-nicotinic acetylcholine receptor availability and are incentivized for successfully abstaining from cigarettes for up to 8 days.
  [F18]-ASEM (3-(1,4-diazabicyclo[3.2.2]nonan-4-yl)-6-[18F]fluorodibenzo[b,d]thiophene 5,5-dioxide): Brain imaging of alpha-7 nicotinic acetylcholine receptors
  Contingency Management: Incentive payments contingent upon provision of samples that meet criterion levels of exhaled carbon oxide and urinary cotinine at study visits
Period: Overall Study
Arm/Group | Tobacco Smokers During a Quit Attempt
Started | 15
Completed | 3
Not Completed | 12

BASELINE CHARACTERISTICS:
Groups:
- Tobacco Smokers During a Quit Attempt: Abstinent tobacco smokers receiving a MRI and a PET scan with the alpha7-nAChR radiotracer [18F]-ASEM to assess alpha-7-nicotinic acetylcholine receptor availability and are incentivized for successfully abstaining from cigarettes for up to 8 days.
  [F18]-ASEM (3-(1,4-diazabicyclo[3.2.2]nonan-4-yl)-6-[18F]fluorodibenzo[b,d]thiophene 5,5-dioxide): Brain imaging of alpha-7 nicotinic acetylcholine receptors
  Contingency Management: Incentive payments contingent upon provision of samples that meet criterion levels of exhaled carbon oxide and urinary cotinine at study visits
Arm/Group | Tobacco Smokers During a Quit Attempt
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36 (5.257)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Cigarettes per day at intake [Mean (Standard Deviation); unit: Cigarettes per day] | 15.875 (4.673)

OUTCOME MEASURES:

1. Primary Outcome: Distribution Volume (VT) as Determined by [18F]-ASEM PET Scan
Description: Distribution volume (VT) in volumes of interest (VOI) in tobacco smokers. VOI are cingulate, hippocampus, frontal cortex, amygdala, and ventral striatum. VOI are defined via each individual subject's Magnetic Resonance Imaging for anatomical identification of the VOI for alignment with PET images.
Time Frame: 1 day
Population: 3 participants completed this study. No historical controls were matched, data not collected.
Measure: Mean (Standard Deviation); unit: mL/cm^3
Arm/Group | [F18]-ASEM + Contingency Management
Number analyzed (Participants) | 3
mL/cm^3
  Amygdala | 22.640 (1.717)
  Cingulate | 21.588 (2.023)
  Frontal cortex | 22.226 (2.522)
  Hippocampus | 17.431 (0.213)
  Ventral striatum | 20.454 (1.562)

2. Primary Outcome: Total Withdrawal Score on the Minnesota Nicotine Withdrawal Scale (MNWS) on Day of PET Scan
Description: Self-report form has a 15-item list of symptoms where subjects self-rate symptom severity on a scale of 0-4. Validated symptoms for tobacco withdrawal in smokers will be used for the study to quantify total withdrawal symptoms at baseline (smoking as usual), when compared to symptoms on the day of the PET scan. Scores for each item range from 0-4, with 0 representing no symptoms and 4 representing severe withdrawal symptoms. The score range for validated symptoms is 0-36. Higher scores indicate greater nicotine withdrawal severity. Results reported are scores from day of PET scan.
Time Frame: 1 day
Population: Data are from the 3 study completers who completed the PET scan following 1 day of abstinence.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Smokers During a Quit Attempt
Number analyzed (Participants) | 3
score on a scale | 10.667 (1.528)

3. Primary Outcome: Craving/Urge to Smoke as Determined Via the Questionnaire of Subjective Urges (QSU) on Day of PET Scan
Description: The QSU is a 10-item questionnaire to measure craving/urges to smoke. For each item, subjects rate how strongly the subject feel "right now" on a Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Items are summed to yield two factor scores, Factor 1 Intention/desire to smoke (minimum score=5, maximum score=35), and Factor 2: Relief of negative affect and Urgent desire to smoke (minimum score=5, maximum score=35). Factor 1 and Factor 2 scores are combined, with a score range of 10-70, higher score indicating maximum cravings/urges to smoke (worse). Results reported reflect QSU scores on day of PET scan vs baseline.
Time Frame: 1 day
Population: Study Completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Smokers During a Quit Attempt
Number analyzed (Participants) | 3
score on a scale
  Day of PET | 42.667 (6.429)
  Baseline | 22.7 (1.2)

4. Secondary Outcome: Cigarettes Smoked Per Day
Description: Self-reported number of cigarettes smoked daily using a calendar-based time line method for past 90-days (i.e., time line follow back method) when smoking as usual. Average number of daily cigarettes smoked calculated using past 90 days (3 months).
Time Frame: 3 months
Population: Study Completers
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Arm/Group | Tobacco Smokers During a Quit Attempt
Number analyzed (Participants) | 3
Cigarettes per day | 17.00 (3.00)

5. Secondary Outcome: Number of Days of Smoking Abstinence on Day of PET Scan
Description: Number of days abstinent (collected on day of PET scan) will be determined from counting number of CO-and cotinine-verified abstinence days. Abstinence will be defined as negative breath carbon oxide (CO)6ppm or lower AND urinary cotinine decreased by 25 percent from prior sample or <100 ng/ml.
Time Frame: 1 day
Population: Of the 3 completers all maintained abstinence for 1 day and relapsed to smoking (i.e., has CO above criteria levels) on the day after the pet scan.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tobacco Smokers During a Quit Attempt
Number analyzed (Participants) | 3
Days | 1 (0)

6. Secondary Outcome: Negative Mood as Determined by the Positive and Negative Affect Scale (PANAS)
Description: Consists of two 10-item mood scales to provide independent measures of positive and negative affect. Scores for negative affect subscale when smoking as usual, will be compared to days of CO and/or cotinine verified abstinence. Negative Affect Score: Add the scores on items 2, 4, 6, 7, 8, 11, 13, 15, 18, and 20. Scores can range from 0 - 40, with lower scores representing lower levels of negative affect.
Time Frame: Baseline, Day of PET
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Smokers During a Quit Attempt
Number analyzed (Participants) | 3
score on a scale
  PET day | 4.7 (2.9)
  baseline | 5.7 (1.5)

7. Secondary Outcome: Attention as Assessed by Connors Continuous Performance Task
Description: In this computerized task, a stimuli are presented, and subjects are instructed to respond as fast as possible to a specific target stimuli (X) and refrain from responding to more rarely occurring non-target stimuli (non-X). Inattention is indicated by high numbers of omissions and long reaction times. Omissions result from the failure to respond to target letters (i.e., non-Xs); omissions and reaction times when smoking as usual will be compared to those on visits 1-6 during the quit attempt abstinence days. Higher score for detectability represents worse sustained attention. Score range 0 to 100 with higher score being worse.
Time Frame: Baseline, Day of PET
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Smokers During a Quit Attempt
Number analyzed (Participants) | 3
score on a scale
  Baseline | 43.3 (6.0)
  PET day | 50 (13.5)

8. Secondary Outcome: Performance on the Paced Serial Addition Task (PASAT)
Description: The number of correct responses for each trial of the Paced Serial Addition Task (PASAT); Involves presenting a series of single digit numbers where the two most recent digits must be summed. The participant must respond prior to the presentation of the next digit for a response to be scored as correct. Minimum score is 0 and maximum score is 120, with a lower number representing lower levels of sustained attention.The number of correct responses for each trial (maximum = 60). Data reported are the total (sum) correct responses for 2 trials.
Time Frame: Baseline, Day of PET
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Tobacco Smokers During a Quit Attempt
Number analyzed (Participants) | 3
correct responses
  Baseline | 65.7 (10.5)
  PET day | 71.7 (6.1)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Tobacco Smokers During a Quit Attempt
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT04055467/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT04055467/ICF_001.pdf